CLINICAL TRIAL: NCT05177068
Title: A Phase II Clinical Study of Fruquintinib Combined With Sintilimab and SOX as Conversion Therapy of Potentially Resectable Stage IV Gastric Cancer
Brief Title: Conversion Therapy of Fruquintinib in Combination With Sintilimab and SOX in Unresectable Gastric Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-G103
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — HMPL-013; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): fruquintinib + sintilimab + SOX (S-1 + oxaliplatin)
  Interventions: Drug: fruquintinib + sintilimab + SOX

INTERVENTIONS:
Drug: fruquintinib + sintilimab + SOX — fruquintinib: 4mg/d, qd po, d1-14, q3w; sintilimab: 200 mg/d, IV d1, q3w; S-1: BSA<1.25 m2, 40mg twice/day; BSA1.25-1.5m2, 50mg twice/day; BSA≥1.5 m2, 60mg twice/day, po, d1-14, q3w; oxaliplatin: 130mg/m2, ivgtt 2-6h, d1, q3w

SUMMARY:
This is a phase II study to evaluate the efficacy and safety of combination of fruquintinib (VEGFR 1/2/3 inhibitor), sintilimab (PD-1 inhibitor) and SOX conversion therapy in unresectable advanced gastric cancer patients.

DETAILED DESCRIPTION:
Eligible patients will be given 3 or 6 cycles of combined therapy of fruquintinib + sintilimab + SOX. Then the patients evaluated resectable will be given one additional cycle of combined treatment with sintilimab + SOX, followed by R0 resection. If evaluated unresectable after 6 cycles of combination therapy, the patient will be given palliative first-line treatment. Adjuvant treatment with SOX regimen will be started 4 weeks after R0 resection for a total of 8 cycles in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Signed the Informed Consent Form
* Ages: 18-75 Years (concluding 18 and 75 Years)
* Pathologically confirmed gastric/gastroesophageal junction adenocarcinoma, and meets one of the following conditions: invasion of adjacent organs such as colon, tail of pancreas and spleen; localized peritoneal metastasis; positive exfoliative cytology of ascites; class I, class II, part of class III and very few class IV stage IV gastric adenocarcinoma according to biological behavior; N3; extensive or fused lymph node metastasis; Krukenberg tumor; Liver metastasis limited to one lobe, less than 5cm in diameter, isolated abdominal aortic metastasis, etc;
* Untreated(e.g. radiotherapy, chemotherapy, target therapy and immunotherapy)
* Life expectancy greater than 3 months
* ECOG(Eastern Cooperative Oncology Group) :0~1
* Sufficient organ and bone marrow functions as follows:

  1. Absolute Neutrophil Count (ANC) ≥1.5×109/L, White Blood Cell≥3.5×109/L;
  2. Platelet Count of ≥100×109/L;
  3. Hemoglobin≥90g/L;
  4. Total Bilirubin (TBIL) ≤1.5 x ULN;
  5. ALT and AST<2.5 x ULN, GPT≤1.5×ULN; If there is liver metastasis, then ALT and AST<5.0 x ULN, GPT≤3.0×ULN;
  6. Serum Creatinine (SCr) ≤1.0×ULN;
  7. Endogenous creatinine clearance rate > 60ml / min (Cockcroft Gault formula);
* No severe dysfunction of heart, lung and liver; No jaundice and gastrointestinal obstruction; No acute infection
* Not participating in other clinical trials 4 weeks before and during the treatment

Exclusion Criteria:

* Known HER-2 positive
* Distal metastasis to lung, brain, and bone
* Have received operation on the stomach
* A history of other malignancies within 5 years prior to inclusion, except for cervical carcinoma in situ, basal or squamous cell skin cancer
* Patients with any active autoimmune disease or a documented history of autoimmune disease within 4 weeks prior to enrollment
* Previously received allogeneic bone marrow transplantation or organ transplantation
* Known hypersensitivity to any of the study drugs or excipients
* Hypertension that is not controlled by the drug, and is defined as: SBP ≥150 mmHg and/or DBP ≥90 mmHg
* International normalized ratio (INR) > 1.5 or partially activated prothrombin time (APTT) > 1.5 × ULN
* Poorly controlled diabetes before enrollment
* Clinically significant electrolyte abnormalities judged by researchers
* With any diseases or conditions that affected drug absorption, or the patient could not take drugs orally
* Patients with obvious evidence of bleeding tendency or medical history within 3 months before enrollment, hemoptysis or thromboembolism within 12 months
* Cardiovascular diseases with significant clinical significance, including but not limited to acute myocardial infarction, severe / unstable angina pectoris or coronary artery bypass grafting within 6 months before enrollment; Congestive heart failure, New York Heart Association (NYHA) grade > 2; ventricular arrhythmia requiring drug treatment; LVEF (left ventricular ejection fraction) < 50%
* Active infection or serious infection that is not controlled by drug (≥CTCAE v5.0 Grade 2）
* History of clinically significant hepatic disease, including, but not limited to, known hepatitis B virus (HBV) infection with HBV DNA positive (copies ≥1×104/ml); known hepatitis C virus infection with HCV RNA positive (copies ≥1×103/m)
* Women who are pregnant or lactating
* Urinary protein ≥ ++, and the 24-hour urine protein quantification is greater than 1.0 g
* Have any other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other conditions which, according to judgement of the investigator, renders the patient inappropriate for using of the investigational product or may affect interpretation of study results
* Patients considered unsuitable for inclusion in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical complete resection rate (R0) | about 3 years
  This is a complete macroscopic resection of the gross tumor with negative surgical margins

SECONDARY OUTCOMES:
Rate of downstaging | about 3 years
  To determine the rate of downstaging of locally advanced cT3-4 and/or N+ gastric carcinomas after preoperative therapy
Pathological complete response (pCR) rate | about 3 years
  pCR is defined as the absence of residual tumor based on evaluation of the resected esophagogastric specimen according to Becker remission criteria
Major pathological response (MPR) | about 3 years
  MPR is defined as less than 10% residual tumor after neoadjuvant therapy
Objective Response Rate (ORR) | about 3 years
  ORR was defined as the percentage of the participants in the analysis population who had a confirmed CR or PR according to RECIST 1.1 based on investigator assessment.
Event-free survival (EFS) | about 3 years
  Event-free survival (EFS) is defined as the time from treatment initiation until the occurrence of any predefined event, including disease progression preventing planned surgery, local or distant recurrence, or death from any cause.
Overall survival (OS) | about 3 years
  Overall survival (OS) [time frame: from the initial date of neoadjuvant therapy to the date of death due to any cause. Patients without documentation of death at the time of analysis will be censored at the last follow-up date]. Estimated using Kaplan-Meier method.
adverse event (AEs) | about 3 years
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
R0 Surgical Conversion Rate | about 3 years
  R0 Surgical Conversion Rate is defined as the proportion of R0 resections among patients who completed planned conversion therapy and underwent surgical exploration.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Tumor Hospital, Zhengzhou, Henan, China